CLINICAL TRIAL: NCT00265252
Title: Alendronate in the Prevention of Collapse of Femoral Head in Non-Traumatic Osteonecrosis
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Kaohsiung Medical University Chung-Ho Memorial Hospital (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry); National Cheng-Kung University Hospital (Other); National Taiwan University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: fosamax 01
Record Dates: First submitted 2005-12-12; First posted 2005-12-14 (Estimated); Last update posted 2008-02-27 (Estimated); Status verified 2007-04

CONDITIONS: Non-Traumatic Osteonecrosis
Keywords: osteonecrosis; total hip replacement
MeSH Terms: conditions — Osteonecrosis | interventions — Alendronate

INTERVENTIONS:
Drug: Alendronate

SUMMARY:
To determine the cumulative incidence of total hip replacement, time to event after treatment with Fosamax or placebo during the study peroid

DETAILED DESCRIPTION:
To determine the cumulative incidence of total hip replacement and collpase of femoral head, time to event after treatment with Fosamax or placebo during the study peroid

ELIGIBILITY:
Inclusion Criteria:

* osteonecrosis of femoral head
* be able to provide singed informed consent

Exclusion Criteria:

* prior bisphosphonate use
* pregnant or lactating woman
* bilateral hip replacement

Ages: 20 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60
Dates: Start 2005-06; Study Completion 2008-06 (Estimated)

PRIMARY OUTCOMES:
the cumulative of total hip replacement

SECONDARY OUTCOMES:
necrotic area
Harris hip score

CONTACTS AND LOCATIONS:
Overall Officials: Gwo-Jaw Wang, MD, Study Chair — Kaohsiung Medical University
Locations (1):
- Kaohsiung Medical University Chung-Ho Memorial Hospital, Kaohsiung City, Taiwan

REFERENCES:
- [Background] Lai KA, Shen WJ, Yang CY, Shao CJ, Hsu JT, Lin RM. The use of alendronate to prevent early collapse of the femoral head in patients with nontraumatic osteonecrosis. A randomized clinical study. J Bone Joint Surg Am. 2005 Oct;87(10):2155-9. doi: 10.2106/JBJS.D.02959. PMID 16203877
- [Derived] Chen CH, Chang JK, Lai KA, Hou SM, Chang CH, Wang GJ. Alendronate in the prevention of collapse of the femoral head in nontraumatic osteonecrosis: a two-year multicenter, prospective, randomized, double-blind, placebo-controlled study. Arthritis Rheum. 2012 May;64(5):1572-8. doi: 10.1002/art.33498. PMID 22127729